CLINICAL TRIAL: NCT06328699
Title: Randomized Pilot Study of Chaplain-Delivered Compassion Meditation for Patients Receiving Stem Cell Transplantation
Brief Title: Chaplain-Delivered Compassion Meditation to Improve Spiritual Care of Patients Receiving Stem Cell Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jennifer Mascaro, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006456; EU6011-23 (Other: Emory University Hospital/Winship Cancer Institute); K01AT010488 (NIH); P30CA138292 (NIH)
Record Dates: First submitted 2023-12-04; First posted 2024-03-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Spiritual Therapies; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Chaplain delivered compassion meditation) (Experimental): Patients receive chaplain led compassionate centered spiritual health sessions over 30 minutes, twice per week for up to 2 weeks.
  Interventions: Procedure: Spiritual Therapy
- Arm II (Traditional chaplain consultation) (Active Comparator): Patients receive a traditional chaplain consultation and care upon request, per standard of care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Procedure: Spiritual Therapy — Undergo chaplain led compassionate centered spiritual health sessions
  Arms: Arm I (Chaplain delivered compassion meditation)
Other: Best Practice — Receive a traditional chaplain consultation and will receive care upon request
  Other Names: best practice, standard of care, standard of care, standard therapy
  Arms: Arm II (Traditional chaplain consultation)

SUMMARY:
This clinical trial tests the feasibility, implementation and acceptability of chaplain delivered compassion meditation in order to improve spiritual care for patients receiving stem cell transplantation. Hospital chaplains play a vital role in delivering emotional and spiritual care to a broad range of both religious and non-religious patients for a wide variety of stressors, and extensive research indicates that spiritual consults impact patient outcomes and satisfaction. Compassion meditation is a secularized, research-based mindfulness and compassion meditation program designed to expand and strengthen compassion for self and others. Practices include training in attentional stability and increased emotional awareness, as well as targeted reflections to appreciate one's relationship with self and others. By centering the mind, controlling debilitating ruminative thoughts, and cultivating personal resiliency and an inclusive and more accurate understanding of others. Engaging in chaplain delivered compassion meditation may improve the spiritual care for patients receiving stem cell transplantation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the feasibility, adoption, extent of implementation, acceptability and fidelity of chaplain-delivered compassion-centered spiritual health (CCSH).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive chaplain-led compassionate centered spiritual health sessions over 30 minutes, twice per week for up to 2 weeks.

ARM II: Patients receive a traditional chaplain consultation and care upon request, per standard of care.

After completion of study treatment, patients are followed up at 80-100 days and 6 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: Within 6 weeks of scheduled hematopoietic stem cell transplant (HSCT)
* PATIENT: > 18 years of age
* PATIENT: Speak and read English
* CHAPLAIN: Emory Healthcare chaplain

Exclusion Criteria:

* PATIENT: Patients will be excluded if they are cognitively impaired, on a ventilator, or are in a room requiring enteric precautions or airborne precautions (e.g., use of an N-95 mask requiring fit-testing) to enter
* CHAPLAIN: There will be no exclusion criteria and no consequence to the chaplains for refusing to volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility - patient enrollment and treatment-specific retention rates | Up to 8 months
  Will measure and characterize the proportion of eligible patient screens who enroll and treatment-specific retention rates.

SECONDARY OUTCOMES:
Patient Characteristics Affecting Acceptability - Chaplain Satisfaction Survey | Up to 8 months
  We will examine whether scores on the chaplain satisfaction survey vary based on patient sociodemographic variables (biological sex, race)
Functional Assessment of Cancer Therapy-Bone Marrow Transplant [FACT-BMT] | Up to 8 months
  Impact of chaplain-delivered compassion-centered spiritual health on quality of life
Acceptability - Chaplain Satisfaction Survey | Up to 8 months
  Will administer a post- chaplain-based compassion treatment (CBCT) intervention using chaplain satisfaction survey and will ask patients after each session if they would like to continue receiving CBCT sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States